CLINICAL TRIAL: NCT00921492
Title: Does Low-frequency Electro-acupuncture Restore Sensitivity of the Gonadotropin-releasing Hormone Pulse Generator and Stress Axis in Polycystic Ovary Syndrome
Brief Title: Acupuncture and Gonadotropin-releasing Hormone Pulse Generator and Stress Axis in Polycystic Ovary Syndrome
Acronym: PCOSLFEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCOSLFEA-17611; 2008-72VP-15445-01A; ALFFGBG-10984
Record Dates: First submitted 2009-06-12; First posted 2009-06-16 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Luteinizing hormone; Cortisol; HPA axis; HPO axis; Ovulation; Heart rate variability; Psychological distress and quality of life
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-frequency electro-acupuncture (Experimental)
  Interventions: Device: Low-frequency electro-acupuncture (EA)
- Meeting a therapist - attention (Active Comparator)
  Interventions: Other: Meeting a therapist - attention control

INTERVENTIONS:
Device: Low-frequency electro-acupuncture (EA) — 2 Hz EA during 30 minutes, twice a week, 14 weeks.
  Arms: Low-frequency electro-acupuncture
Other: Meeting a therapist - attention control — Meeting a therapist, twice a week during 30 minutes in order to control for the increased amount of attention.
  Arms: Meeting a therapist - attention

SUMMARY:
Hypothesis The overall hypothesis is that non-obese (BMI <30) women with PCOS have high luteinising hormone (LH) and cortisol pulse frequency and amplitude and that repeated low-frequency EA restore these alterations and induce ovulation.

DETAILED DESCRIPTION:
Aim 1. Elucidate if low-frequency EA induce ovulation and restore LH frequency and amplitude as well as sex steroid secretion as compared to a control group receiving same amount of attention.

Aim 2. Elucidate if low-frequency EA restore cortisol frequency and amplitude compared to a control group receiving same amount of attention.

Aim 3. Elucidate if low-frequency EA restore psychological distress and quality of life as compared to a control group receiving same amount of attention.in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 39 years, inclusive
* 30 ≤ BMI
* History of irregular menstrual cycles
* Clinical and/or biochemical androgen excess (determined during screening)

Exclusion Criteria:

Medical Exclusion Criteria

* History or clinical manifestation of; cardiovascular disease, diabetes (Type 1 or Type 2), any other significant endocrine or metabolic disorder.
* Regular use of medications for weight control, psychosis and thyroid disease. A 3 month washout period will be permitted for contraceptives.

Psychiatric and Behavioral Exclusion Criteria

* Pregnant or breast-feeding women

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Frequent blood sampling every 10th minute during an overnight stay in order to measure changes in LH and cortisol pulsatility before and after treatment. A third assessment will be made in those participants who ovulate during the 14 week study. | 16 weeks

SECONDARY OUTCOMES:
Ovulation, health related quality of life | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Neuroscience and Physiology, Sahlgrenska Academy, Göteborg University, Gothenburg, Sweden

REFERENCES:
- [Derived] Johansson J, Redman L, Veldhuis PP, Sazonova A, Labrie F, Holm G, Johannsson G, Stener-Victorin E. Acupuncture for ovulation induction in polycystic ovary syndrome: a randomized controlled trial. Am J Physiol Endocrinol Metab. 2013 May 1;304(9):E934-43. doi: 10.1152/ajpendo.00039.2013. Epub 2013 Mar 12. PMID 23482444